CLINICAL TRIAL: NCT05542082
Title: OUS Multicenter Pilot Study of the CHILLS Cryotherapy System for the Treatment of Obstructive Sleep Apnea (ARCTIC-2)
Brief Title: Pilot Study of the CHILLS Cryotherapy System for the Treatment of OSA
Acronym: ARCTIC-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Cryosa elected to terminate the study and discontinue further follow-up after all willing and available subjects had completed the 6-month follow-up. The primary endpoint of 90-days of follow up was met for all active subjects.
Sponsor: Cryosa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10721
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental): CHILLS Procedure
  Interventions: Device: CHILLS Procedure

INTERVENTIONS:
Device: CHILLS Procedure — Cryotherapy

SUMMARY:
This is a prospective, multicenter, non-randomized single-arm safety and efficacy study to:

* Collect data to evaluate the safety of CHILLS cryotherapy to treat OSA in patients with moderate to severe disease.
* Evaluate the chronic performance of the CHILLS system and collect clinical measures for therapy effectiveness that will be used to demonstrate safety and effectiveness in the next clinical study.

DETAILED DESCRIPTION:
The study will enroll up to 3 sites in Latin America, enrollment is competitive.

Up to 70 subjects will receive treatment and be followed through their 3-month visit.

Long-term follow-up will continue every 6 months out to 2 years post-procedure, with an option to follow patients up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

Likely suffer moderate to severe OSA based on history and physical or have an established diagnosis of moderate to severe OSA (AHI ≥ 10) based on a prior sleep study.

A confirmation baseline sleep study will be performed after enrollment to verify AHI ≥ 10 and ≤ 50, and mixed and central apneas total ≤ 25% of apneas for continued eligibility.

Have either failed Positive Airway Pressure (PAP) therapy or decline PAP therapy

BMI of 25 - 40 kg/m2 at enrollment

Negative result for COVID-19 polymerase chain reaction (RT-PCR) test and absence of clinical symptoms for long COVID-19 relating to deterioration of taste, smell.

Exclusion Criteria:

Unable or incapable of providing informed written consent

Unwilling or incapable of returning to all follow-up visits and sleep studies, including evaluation procedures and filling out questionnaires

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Procedure-Related Complications | 90 Days
  No serious procedure-related complications including death; loss of the airway requiring post-anesthesia care unit (PACU) re-intubation; persistent loss (more than 30 days) of tongue movement; bleeding requiring surgical intervention or transfusion; device- or procedure-related hospital re-admission; or De novo clinically significant hypoxemia (immediate or delayed) with SpO2 < 70% for > 10% of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Rowley, MD, Principal Investigator — San Fernando Specialized Center
Locations (2):
- Panama (2):
  - Punta Pacifica Hospital, Panama City, Provincia de Panamá
  - Paitilla Medical Center, Panama City

IPD SHARING:
Plan to Share IPD: No